CLINICAL TRIAL: NCT01662687
Title: Randomized Study of the Efficacy and Safety of Transdermal Granisetron Compared With Intravenous and Oral Agent in the Control of Nausea and Vomiting Induced by Moderately Emetogenic Chemotherapy
Brief Title: Phase 4 Trial to Evaluate the Efficacy and Safety of Sancuso Patch in CINV (Chemotherapy-induced Nausea and Vomiting) Associated With the Administration of MEC (Moderately Emetogenic Chemotherapy)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LG-SCSCL002
Record Dates: First submitted 2012-08-08; First posted 2012-08-10 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Chemotherapy-induced Acute or Delayed Nausea and Vomiting (CINV)
MeSH Terms: conditions — Vomiting

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sancuso patch (Experimental)
  Interventions: Drug: Sancuso patch
- Kytril (Active Comparator)
  Interventions: Drug: Kytril inj.+Kytril tab.

INTERVENTIONS:
Drug: Sancuso patch — Eligible patients were randomized to Sancuso patch or Kytril groups and received the assigned treatment for 4days.
  Experimental arm: Sancuso patch (34.3mg) applied to upper, outer arm 2days (48-24 hours) prior to start of chemotherapy.
  Arms: Sancuso patch
Drug: Kytril inj.+Kytril tab. — Eligible patients were randomized to Sancuso patch or Kytril groups and received the assigned treatment for 4days.
  Active Comparator arm:
  * Kytril inj. 3mg: administered by intravenous infusion at least 5 minutes, just before the first chemotherapy (Day 1).
  * Kytril tab. 1mg: administered twice a day by orally at Day 2~4.
  Arms: Kytril

SUMMARY:
Multicenter, randomized, open-label, paralled-group, active-controlled study. The study is to demonstrate non-inferiority of the Granisetron Transdermal Delivery System (GTDS) compared with the intravenous and oral Granisetron in the prevention of CINV associated with moderately emetogenic Chemotherapy.

Patients scheduled to receive the one cycle of a ME chemotherapy regimen administered for 1-4 days will attend a Screening Visit 2 to 28 days before start of ME chemotherapy. Eligible patients will be randomized to 1 of 2 treatment groups at the Randomization Visit (1 to 2 days prior to ME chemotherapy).

* Sancuso patch
* Kytril inj.+Kytril tab.

The patch will be applied 2days (48-24h) prior to first daily dose of the moderately emetogenic chemotherapy regimen and remain in place for 6 days. The patient will be assessed daily until 4days after first chemotherapy administration. Adverse Events (AEs) will be collected until 14 days after the final dose of IP. Non-serious AEs will be followed-up until 14 days after the final dose of IP. Serious adverse events will be followed-up until they are resolved, stable or until the patient is lost to follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged over 20 yrs
2. Histologically and/or cytologically proven cancer patients
3. Eastern Cooperative Oncology Group performance status 0, 1, 2
4. A cycle of moderately emetogenic chemotherapy(NCCN Guidelines)
5. Life expectancy of ≥ 3 months
6. Normal liver function and renal function(total bilirubin ≤ 1.5 ULN, AST/ALT ≤ 2.5 ULN, in case of liver metastases AST/ALT ≤ 5 ULN, serum creatinine ≤ 1.5 ULN) patients
7. Patients who signed the informed consent form

Exclusion Criteria:

A. Previous History

1. Hypersensitivity to adhesive plasters
2. Contraindications to 5-HT3 receptor antagonists
3. Any other relevant medical history (at the discretion of the investigator)

B. Concomitant Medical Condition

1. Current alcohol, drug or medication abuse
2. Currently pregnant or breast feeding women, including planning pregnancy
3. Clinically relevant abnormal laboratory values (at the discretion of the investigator)
4. Clinically relevant heart, hepatic, renal, infectious, neurological or psychiatric disorders, or any other major systemic illness (at the discretion of the investigator)
5. Any cause for nausea and vomiting other than CINV
6. Any episode of retching, vomiting or uncontrolled nausea in the 72 h period prior to the chemotherapy administration
7. Clinically relevant abnormal ECG parameters (at the discretion of the investigator)

C. Concomitant Therapy/Medication

1. Concomitant radiotherapy of total body, brain or upper abdomen within one week prior to the study entry or planned during the study
2. Intake of medication to control the symptoms of a brain tumor, brain metastasis or seizure disorder or neuropathy (unless peripheral neuropathy at the discretion of the investigator)
3. Patients using selective serotonin reuptake inhibitor (SSRI) antidepressants (unless a stable dose for the duration of the study)
4. Receipt of a narcotic analgesics (acceptable at the discretion of the investigator)
5. Receipt of any other clinical trial drug < 30 days before the study or during the study
6. Scheduled to receive a neurokinin NK1 receptor antagonist, dopamine receptor antagonist or another 5-HT3 receptor antagonist at 72 h prior to the administration of the chemotherapy or scheduled to do those medication during chemotherapy duration
7. Drugs known to increase the QTc interval (unless a stable dose for the duration of the study at the discretion of the investigator)

D. Other

1. Patients unlikely to comply with the study protocol (at the discretion of the investigator), e.g. uncooperative attitude, inability to return for follow-up visits and unlikelihood of completing the study
2. The patch adhesion level was not more than 50% on the day of chemotherapy or the patch was not attached within two days before the chemotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Estimated)
Dates: Start 2012-02; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
The percentage of patients achieving Complete Response (CR) without rescue therapy from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen

SECONDARY OUTCOMES:
The percentage of patients achieving Complete Response (CR) | overall (Day 1~4)
The percentage of patients achieving Complete Control (CC) without rescue therapy from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen
The percentage of patients achieving Complete Control (CC) | overall (Day 1~4)
severity of nausea | overall (Day 1~4)
severity of vomiting | overall (Day 1~4)
Frequency of nausea from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen
Frequency of vomiting from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen | from the first administration until 24h after the start of the last day's administration of the ME chemotherapy regimen
Patient's satisfaction with anti-emetic therapy (Changes from Baseline to Day 5) | from baseline to Day 5
  The patient's response to anti-emetic therapy was assessed and recorded by patients at Visit 3 (Baseline) and Visit 7 (Day 5). The patient was asked to evaluate his/her satisfaction with the control of nausea and vomiting by marking the FLI-E (Functional Living Index - Emesis) with vertical lines.
The percentage of patients achieving Complete Response (CR) | per day (Day 1, 2, 3, 4)
The percentage of patients achieving Complete Control (CC) | per day (Day 1, 2, 3, 4)
severity of nausea | per day (Day 1, 2, 3, 4)
severity of vomiting | per day (Day 1, 2, 3, 4)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Seok Ahn, MD, PhD, Principal Investigator — Samsung Medical Center; Tae Won Kim, MD, PhD, Principal Investigator — Asan Medical Center; Dong Bok Shin, MD, PhD, Principal Investigator — Gachon University Gil Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim JE, Hong YS, Lee JL, Kim KP, Park SJ, Sym SJ, Shin DB, Lee J, Park YS, Ahn JS, Kim TW. A randomized study of the efficacy and safety of transdermal granisetron in the control of nausea and vomiting induced by moderately emetogenic chemotherapy in Korean patients. Support Care Cancer. 2015 Jun;23(6):1769-77. doi: 10.1007/s00520-014-2507-6. Epub 2014 Dec 3. PMID 25465680